CLINICAL TRIAL: NCT03438500
Title: The Impact of Cardiac Shock Wave Treatment in Patients With Reduced Coronary Flow Reserve in the Absence of Epicardial Coronary Artery Stenoses: A Pilot Study
Brief Title: Cardiac Shock Wave Treatment in Patients With Reduced Coronary Flow Reserve
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Sponsor & PI decision
Sponsor: Storz Medical AG (Industry)
Collaborators: Technical University of Munich (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CSW-1814-SCH-0010-S
Record Dates: First submitted 2018-02-12; First posted 2018-02-19 (Actual); Last update posted 2022-10-31 (Actual); Status verified 2022-10

CONDITIONS: Refractory Angina Pectoris; Ischemic Heart Disease; Coronary Artery Disease
MeSH Terms: conditions — Angina Pectoris; Myocardial Ischemia; Coronary Artery Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Active Shockwave Therapy (Experimental): Patients in this group receive shockwave therapy.
  Interventions: Device: Cardiac Extracorporeal Shockwave Therapy (Modulith SLC)

INTERVENTIONS:
Device: Cardiac Extracorporeal Shockwave Therapy (Modulith SLC) — 40 - 60 spots per visit (200 shots/spot) at Energy Level 3
  Other Names: Modulith SLC; Extracorporeal Cardiac Shockwave Therapy (CSWT)

SUMMARY:
The purpose of the study is to assess the feasibility of Cardiac Shock Wave Treatment in patients with anginal chest pain and evidence of abnormal myocardial perfusion under stress in the absence of significant stenoses of the epicardial coronary arteries.

DETAILED DESCRIPTION:
This is a mono-center, prospective, single arm, pilot study designed to assess the feasibility of the "Cardiac Shock Wave Treatment" in patients with anginal chest pain and evidence of abnormal myocardial perfusion under stress in the absence of significant stenoses of the epicardial coronary arteries.

A total of 10 subjects will be enrolled in the study. All enrolled study subjects will be assessed for clinical follow-up at the following intervals: 5 and 14 weeks post CSWT procedure.

ELIGIBILITY:
Inclusion Criteria:

* History of anginal chest pain that prompted a myocardial stress test (nuclear myocardial perfusion imaging, stress echocardiography, or perfusion CMR)
* Evidence for stress-induced myocardial ischemia in this examination
* Coronary angiogram showing absence of ≥30% stenosis of epicardial coronary arteries

Exclusion Criteria:

* Participation in other clinical trials
* age <18 years
* Contraindications to under cMRI
* Contraindications to adenosine (severe chronic obstructive pulmonary disease (COPD), asthma, atrioventricular block (AV block) > grade 1)
* Left ventricular thrombus
* Uncontrolled diabetes mellitus
* Uncontrolled arterial hypertension,
* Any other severe chronic illness such as liver or renal failure (glomerular filtration rate (GFR) < 45 ml/min), active neoplastic disease, history of myocardial infarction or coronary revascularization within the past three months
* Patients with pacemaker or implanted cardioverter defibrillator
* Patients after valve surgical replacement
* Patients after interventional valve replacement or reconstruction (e.g. transfemoral aortic valve replacement or MitraClip implantation)
* Pregnancy (a reliable method of contraception must be used for the entire duration of the study)
* Fertile female participants who are capable of bearing children and who do not use a method of contraception that is medically approved by the health authority of the respective country
* Missing capacity to consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2022-09-01 (Estimated); Primary Completion 2022-09-01 (Estimated); Study Completion 2022-09-01 (Estimated)

PRIMARY OUTCOMES:
Change of myocardial perfusion reserve (MPR) | 14 weeks
  Change from baseline in MPR (assessed with quantitative perfusion cardiac magnetic resonance imaging (cMRI)) at 14 weeks
Change of myocardial perfusion reserve (MPR) | 5 weeks
  Change from baseline in MPR (assessed with quantitative perfusion cardiac magnetic resonance imaging (cMRI)) at 5 weeks

SECONDARY OUTCOMES:
Enddiastolic volume | 5 weeks
  Change from baseline in enddiastolic volume (assessed with cMRI and TTE) at 5 weeks
Enddiastolic volume | 14 weeks
  Change from baseline in enddiastolic volume (assessed with cMRI and TTE) at 14 weeks
Endsystolic volume | 5 weeks
  Change from baseline in endsystolic volume (assessed with cMRI and TTE) at 5 weeks
Endsystolic volume | 14 weeks
  Change from baseline in endsystolic volume (assessed with cMRI and TTE) at 14 weeks
Stroke volume | 5 weeks
  Change from baseline in stroke volume (assessed with cMRI and TTE) at 5 weeks
Stroke volume | 14 weeks
  Change from baseline in stroke volume (assessed with cMRI and TTE) at 14 weeks
Ejection fraction | 5 weeks
  Change from baseline in ejection fraction (assessed with cMRI and TTE) at 5 weeks
Ejection fraction | 14 weeks
  Change from baseline in ejection fraction (assessed with cMRI and TTE) at 14 weeks
Regional wall motion | 5 weeks
  Change from baseline in regional wall motion (assessed with steady state free precession cMRI) at 5 weeks
Regional wall motion | 14 weeks
  Change from baseline in regional wall motion (assessed with steady state free precession cMRI) at 14 weeks
Scar extent | 5 weeks
  Change from baseline in scar extent (assessed with late gadolinium enhancement cardiac magnetic resonance imaging (LGE cMRI)) at 5 weeks
Scar extent | 14 weeks
  Change from baseline in scar extent (assessed with late gadolinium enhancement cardiac magnetic resonance imaging (LGE cMRI)) at 14 weeks
Diffuse fibrosis | 5 weeks
  Change from baseline in diffuse fibrosis (assessed with T1 mapping) at 5 weeks
Diffuse fibrosis | 14 weeks
  Change from baseline in diffuse fibrosis (assessed with T1 mapping) at 14 weeks
Severity and frequency of angina | 5 weeks
  Change from baseline in Seattle Angina questionnaire at 5 weeks
Severity and frequency of angina | 14 weeks
  Change from baseline in Seattle Angina questionnaire at 14 weeks
New York Heart Association (NYHA) class | 5 weeks
  Change from baseline in NYHA class at 5 weeks
New York Heart Association (NYHA) class | 14 weeks
  Change from baseline in NYHA class at 14 weeks
Exercise capacity | 5 weeks
  Change from baseline in exercise capacity (assessed by the 6-minute walk test) at 5 weeks
Exercise capacity | 14 weeks
  Change from baseline in exercise capacity (assessed by the 6-minute walk test) at 14 weeks
Quality of life (SF-36) | 5 weeks
  Change from baseline in quality of life (assessed with questionnaire Short Form (SF-36) Health Survey) at 5 weeks
Quality of life (SF-36) | 14 weeks
  Change from baseline in quality of life (assessed with questionnaire Short Form (SF-36) Health Survey) at 14 weeks
New myocardial scarring or fibrotic changes | 5 weeks
  Change from baseline in new myocardial scarring or fibrotic changes (assessed with LGE cMRI) at 5 weeks
New myocardial scarring or fibrotic changes | 14 weeks
  Change from baseline in new myocardial scarring or fibrotic changes (assessed with LGE cMRI) at 14 weeks
Myocardial edema | 5 weeks
  Change from baseline in myocardial edema (assessed with cMRI) at 5 weeks
Myocardial edema | 14 weeks
  Change from baseline in myocardial edema (assessed with cMRI) at 14 weeks
Myocardial hemorrhage | 5 weeks
  Change from baseline in myocardial hemorrhage (assessed with cMRI) at 5 weeks
Myocardial hemorrhage | 14 weeks
  Change from baseline in myocardial hemorrhage (assessed with cMRI) at 14 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Georg Schmidt, Prof. Dr., Principal Investigator — Technische Universität München I. Medizinische Klinik und Poliklinik; Alexander Steger, Dr. med., Principal Investigator — Technische Universität München I. Medizinische Klinik und Poliklinik
Locations (1):
- Technische Universität München I. Medizinische Klinik und Poliklinik, München, Germany

IPD SHARING:
Plan to Share IPD: No